CLINICAL TRIAL: NCT03872037
Title: Selective Dentine Removal in Primary Teeth: a Randomized Clinical Trial
Brief Title: Selective Dentine Removal in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, PhD, Senior Lecturer, Clinical Professor, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLM 7
Record Dates: First submitted 2019-03-04; First posted 2019-03-12 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Caries, Dental
Keywords: minimally invasive dentistry; dental caries; dentine
MeSH Terms: conditions — Dental Caries | interventions — Maxxion

STUDY DESIGN:
Intervention Model Description: A total of 150 children were allocated to two parallel groups: group 1 (G1, n = 70, control, Ketac Molar Easymix®, 3M/ESPE, Seefeld, GE) and group 2 (G2, n = 80, test, Maxxion®, FGM, Joinville, BR). The study was double-blinded, and an operator specialized in paediatric dentistry performed the selective removal of soft dentine and the restoration of the cavity with GIC. During the follow-up periods, the teeth were evaluated via periapical radiography by two trained examiners specialized in radiology. Statistical analysis was performed using Stata 11.2 software (StataCorp, Texas, USA) and a survival curve (Kaplan-Meier).
Who Masked: Participant, Investigator
Masking Description: For the radiographic evaluation, the evaluators had no information about the group to which the parent was randomized. Only the periapical tissues were evaluated, and the coronary portion of the restored tooth was concealed with adhesive tape.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Molars subjected to selective removal and restored with Ketac Molar Easymix
  Interventions: Procedure: Control
- Selective removal of caries and restoration with Maxxion (Experimental): Molars subjected to selective removal and restored with Maxxion
  Interventions: Procedure: Selective removal of carious tissue and restoration with Maxxion

INTERVENTIONS:
Procedure: Selective removal of carious tissue and restoration with Maxxion — Molars subjected to selective removal and restored with Maxxion
  Arms: Selective removal of caries and restoration with Maxxion
Procedure: Control — Molars subjected to selective removal and restored with Ketac Molar Easymix
  Arms: Control

SUMMARY:
Background There is little information regarding the longevity of the restored tooth, considering the health of the pulp-dentine complex, in children who do not sufficiently cooperate with dental treatment.

Aim To evaluate the longevity of primary molar teeth with an occluso-proximal cavity that was treated with the selective removal of carious tissue.

Design A total of 150 children were allocated to two parallel groups: group 1 (G1, n = 70, control, Ketac Molar Easymix®, 3M/ESPE, Seefeld, GE) and group 2 (G2, n = 80, test, Maxxion®, FGM, Joinville, BR). The study was double-blinded, and an operator specialized in paediatric dentistry performed the selective removal of soft dentine and the restoration of the cavity with GIC. During the follow-up periods, the teeth were evaluated via periapical radiography by two trained examiners specialized in radiology. Statistical analysis was performed using Stata 11.2 software (StataCorp, Texas, USA) and a survival curve (Kaplan-Meier).

ELIGIBILITY:
Inclusion Criteria:

* An active denture caries lesion
* The molars in primary, without anterior restoration, with the exclusive involvement of occlusal and mesial or distal surfaces present (International Caries Detection and Evaluation System, ICDAS score 5)

Exclusion Criteria:

* Those who did not accept care after 3 adaptation sessions
* Teeth with the following characteristics were excluded from the study: spontaneous pain, pressure sensitivity, suspected cellulose involvement, necrosis pulp, fistula, or tooth mobility
* Teeth in which extension of the lesion could lead to pulpal exposure were excluded
* Children whose parents or guardians do not sign an Informed Consent Term

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Number of teeth with treatment-related success as assessed by radiographic analysis. | 14-month
  To evaluate the longevity of primary molar teeth with an occluso-proximal cavity that was treated with the selective removal of carious tissue.
Number of teeth with treatment-related success as assessed by radiographic analysis. | 24-month
  To evaluate the longevity of primary molar teeth with an occluso-proximal cavity that was treated with the selective removal of carious tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos P Imparato, PhD, Principal Investigator — Sao Leopoldo Mandic
Locations (1):
- Faculty Sao Leopoldo Mandic, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Priesnitz MC, Celeste RK, Pereira MJ, Pires CA, Feldens CA, Kramer PF. Neighbourhood Determinants of Caries Experience in Preschool Children: A Multilevel Study. Caries Res. 2016;50(5):455-461. doi: 10.1159/000447307. Epub 2016 Aug 17. PMID 27529624
- [Background] Roncalli AG, Sheiham A, Tsakos G, Araujo-Souza GC, Watt RG. Social Factors Associated with the Decline in Caries in Brazilian Children between 1996 and 2010. Caries Res. 2016;50(6):551-559. doi: 10.1159/000442899. Epub 2016 Oct 6. PMID 27705968
- [Background] Hannas AR, Kato MT, Cardoso Cde A, Magalhaes AC, Pereira JC, Tjaderhane L, Buzalaf MA. Preventive effect of toothpastes with MMP inhibitors on human dentine erosion and abrasion in vitro. J Appl Oral Sci. 2016 Jan-Feb;24(1):61-6. doi: 10.1590/1678-775720150289. PMID 27008258
- [Background] Bjørndal L, Ricucci D, 2014. Pulp inflammation: from the reversible inflammation to pulp necrosis during caries progression. In Michel G ed. The Dental Pulp Biology, Pathology, and Regenerative Therapies. Berlin (Germany): Springer. pp 125-139.
- [Background] Banerjee A, Domejean S. The contemporary approach to tooth preservation: minimum intervention (MI) caries management in general practice. Prim Dent J. 2013 Jul;2(3):30-7. doi: 10.1308/205016813807440119. PMID 24340496
- [Background] Baelum V, Hintze H, Wenzel A, Danielsen B, Nyvad B. Implications of caries diagnostic strategies for clinical management decisions. Community Dent Oral Epidemiol. 2012 Jun;40(3):257-66. doi: 10.1111/j.1600-0528.2011.00655.x. Epub 2011 Nov 21. PMID 22103270
- [Background] Calvo AF, Kicuti A, Tedesco TK, Braga MM, Raggio DP. Evaluation of the relationship between the cost and properties of glass ionomer cements indicated for atraumatic restorative treatment. Braz Oral Res. 2016;30:S1806-83242016000100201. doi: 10.1590/1807-3107BOR-2016.vol30.0008. Epub 2015 Dec 15. PMID 26676191